CLINICAL TRIAL: NCT03657121
Title: COPD: Comparison of Existing Prognostic Tools for 1 Year Mortality and Assessment of Symptom Burden to Facilitate Advance Care Planning
Brief Title: Mortality and Symptom Burden Post Hospitalisation With COPD
Acronym: MoSHCOPD
Status: Completed | Type: Observational
Sponsor: Northumbria Healthcare NHS Foundation Trust (Other)
Collaborators: National Institute for Health Research, United Kingdom (Other Government); Newcastle-upon-Tyne Hospitals NHS Trust (Other); Hospice UK (Unknown)
Responsible Party: Principal Investigator, Sarah Gillespie, Respiratory Palliative Care Fellow, Northumbria Healthcare NHS Foundation Trust
Other Study IDs: 244285
Record Dates: First submitted 2018-08-02; First posted 2018-09-04 (Actual); Last update posted 2021-03-03 (Actual); Status verified 2021-03

CONDITIONS: Pulmonary Disease, Chronic Obstructive; Pulmonary Disease, Obstructive; Emphysema; Chronic Bronchitis; Chronic Bronchitis With Airways Obstruction; Chronic Bronchitis With Acute Exacerbation
Keywords: Prognosis; Palliative Care; End Stage; Mortality; Palliative; Advance Care Planning; Symptom; Exacerbation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Diseases, Obstructive; Emphysema; Bronchitis, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Chronic Obstructive Pulmonary Disease (COPD) is a common progressive lung disease which causes breathlessness and frequent exacerbations, with patients often requiring hospitalisation. Patients with severe COPD commonly become housebound and lose their independence. They have a higher symptom burden than those with incurable lung cancer, yet are less likely to receive specialist palliative care, or to have been engaged in advance care planning (where patients discuss and often document their wishes regarding their future care). Hospital admissions become increasingly common towards the end-of-life; therefore, hospitalisation is a good opportunity to identify patients at risk of poor outcome. Such patients may wish to consider alternatives to admission and avoid intrusive treatments. Unfortunately, predicting which patients are likely to die in the near future is challenging thus far.

The first step required to improve provision of palliative care services, and ensure patients are given the opportunity to make truly informed decisions about their future care, is accurate identification of those most likely to benefit.

Well-designed clinical (prognostic) tools outperform clinician judgement in most settings. The investigators will compare the accuracy of one year mortality prediction of several clinical tools in patients who survive a COPD exacerbation requiring admission. This will initially be performed using existing data collected during previous research (the 1,593 patient validation study for the PEARL score - Previous admissions, extended Medical Research Council Dyspnoea score, Age, Right and Left heart failure), then confirmed in at least 310 patients admitted uniquely and consecutively with an exacerbation of COPD. The latter group of patients will be invited to participate in a longitudinal follow-up study, assessing symptom burden, quality of life, and readmissions over one year.

DETAILED DESCRIPTION:
The PEARL (Previous admissions, Extended Medical Research Council Dyspnoea Score, Age, Right-sided heart failure and Left-sided heart failure) score predicts readmission or death within 90 days of discharge following an exacerbation of Chronic Obstructive Pulmonary Disease (ECOPD), and was developed by the lead supervisor's research team. Within the PEARL derivation cohort (2 hospitals, 824 patients), they have developed a novel tool to predict one year survival. The performance of this novel tool and existing Chronic Obstructive Pulmonary Disease (COPD) prognostic tools will be compared in the PEARL validation cohort (6 hospitals, 1,593 patients). The existing tools are the Body Mass Index, Airflow Obstruction, Dyspnoea and Exacerbations (BODEX) index (score range 0-9); PEARL score (score range 0-9); COPD Gold Standards Framework Prognostic Indicator Guidance (COPD PIG); Comorbidity, Obstruction, Dyspnoea and Exacerbations (CODEX) index (score range 0-10); Age, Dyspnoea and Obstruction (ADO) index (score range 0-14); Dyspnoea, Obstruction, Smoking, Exacerbation (DOSE) index (score range 0-8), the Supportive and Palliative Care Indicators Tool (SPICT) and another tool recently developed by another centre (PubMed reference not yet available). COPD-PIG and SPICT are not scored in the same manner and therefore do not have a range.

Performance of all tools will also be further prospectively assessed in a minimum of 310 patients. The COPD-PIG is intended to only be scored in patients who the clinician "would not be surprised" if they died within one year; the performance of this tool cannot be fully assessed retrospectively. Prospective validation will also allow an assessment of the ease of data collection; this is not available for the existing PEARL cohort but is a key consideration in selection of the final tool to ensure it is appropriate for widespread use on hospital wards. Consecutive, unique patients admitted to Northumbria Healthcare NHS Foundation Trust and Newcastle Upon Tyne Hospitals NHS Foundation Trust with ECOPD will be identified. Demographic and clinical indices, including the components of the nine prognostic tools, will be collected. Caldicott and ethics committee approval are in place (REC:18/NE/0226). Hospital readmissions, utilisation of other healthcare services such as the local palliative care teams and Hospice and survival will be assessed over one year. In common with similar studies, this validation study will be non-consenting.

Patients identified as high-risk by the selected tool who survive beyond one year may still warrant palliative care input if their symptom burden is high. The patients enrolled in the validation study will be invited to participate in a consenting longitudinal outcomes study, aiming for at least 50% participation. Symptom burden and functional status will be assessed using the St George's Respiratory Questionnaire (SGRQ), Hospital Anxiety and Depression Score (HADS), Australian modified Karnofsky Score (AKPS), Extended Medical Research Council Dyspnoea (eMRCD) score, and modified Borg scale at baseline, and 1, 3, 6 and 12 months. The baseline and 3 month assessments will be conducted via face to face meetings. The additional 1, 6 and 12 month assessments will be conducted over the phone. This data will be used both to calculate the relationship between symptom burden and death, and to identify the characteristics of patients who are especially symptomatic.

The characteristics of the cohort will be summarised using standard descriptive statistics appropriate to the level and distribution of the data. Groups will be compared (including by mortality outcome) using standard tests of statistical inference (e.g. t-test, Mann-Whitney U test, Fishers exact test). The performance of candidate prognostic tools will be compared by 1) assessing the positive and negative predictive value within the high-risk and low risk groups respectively; and 2) Area Under the curve of the Receiver Operating Characteristic (AUROC) analysis, with performance compared using the method of DeLong et al. Where data imputation is required, this will be done using multiple imputation methods. Statistical significance will be set at 5% throughout. The statistical analysis plan will be finalised prior to end of recruitment to avoid potential bias.

ELIGIBILITY:
Inclusion Criteria:

1. Age 35 years or older.
2. Smoking history greater than or equal to 10 pack years.
3. Obstructive spirometry (FEV1/FVC < 0.7).
4. ECOPD primary diagnosis.
5. Survival to discharge.

Exclusion Criteria:

1. Previous inclusion in the study.
2. Malignant neoplasm or other pathology likely to limit survival to less than 1 year.
3. For the longitudinal study only, inability to give informed consent.

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive, unique patients admitted to Northumbria Healthcare NHS Foundation Trust or Newcastle Upon Tyne Hospitals NHS Foundation Trust with an exacerbation of Chronic Obstructive Pulmonary Disease (ECOPD) will be identified and included in the non consenting prognostic study. All eligible patients within this group will be approached to participate in the longitudinal study and will only be included if they consent to do so.
Sampling Method: Probability Sample
Enrollment: 447 (Actual)
Dates: Start 2019-01-16 (Actual); Primary Completion 2020-12-18 (Actual); Study Completion 2020-12-18 (Actual)

PRIMARY OUTCOMES:
Positive predictive value of the prognostic tools listed for prediction of one year mortality. | 12 months
  This is an exploratory study. The optimal tool to identify patients for advance care planning needs to offer high PPV (i.e. the substantial majority of those identified at high risk of dying should not survive beyond one year) and reasonably high sensitivity (i.e. most deaths within one year should be identified). Ease of completion must also be considered as this will strongly influence engagement.
Sensitivity of the prognostic tools listed for prediction of one year mortality. | 12 months
  As above

SECONDARY OUTCOMES:
Ease of completion of prognostic tools assessed by Likert scale | 12 months
  Commonly used psychometric scale, which will be utilised by the principal investigator to score the practical ease of completion of the prognostic tools for individual patients. A 10 point scale (score range 1-10) will be utilised with higher numbers conferring greater ease.
Ease of completion of prognostic tools assessed by missing data. | 12 months
For each prognostic tool, the area under the receiver operating characteristic curve. | 12 months
Negative predictive value of the prognostic tools for prediction of one year mortality. | 12 months
Hospital readmission rates at 30, 90 and 365 days. | 12 months
Proportion of patients on the palliative care register and relation to mortality. | 12 months
Utilisation of palliative care services: hospice; community palliative care team. | 12 months
  Rates of usage of these services will be identified at 12 months
Inter-observer agreement on scoring of the prognostic tools | 12 months
  A random sample of patients will be selected and the prognostic tools re-scored by a different member of the research team to identify disagreements.
Determine baseline St George's Respiratory Questionnaire score | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools.
  SGRQ is a validated questionnaire which measures the health status of patients with COPD, with a score ranging from 0 (no impairment) to 100 (worst possible health). Patients in a high mortality risk group identified for advance care planning who do not die are not "false positives" if they have a high symptom burden. The proportion of patients with high symptom burden not identified is also clinically relevant. This and the subsequent secondary outcomes are therefore important in this regard.
Determine baseline Hospital Anxiety and Depression Score | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Determine baseline modified Borg score | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. The modified Borg scale is validated to assess breathlessness and is scored from 0 (not breathless) to 10 (maximal breathlessness).
Assess baseline Australia-modified Karnofsky Performance Status | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. AKPS is a validated 10 point scale measuring performance status with 0 being normal health and 100 being dead.
Mean change in SGRQ compared to MCID. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. MCID is the minimal clinically important difference for the validated tool. SGRQ is a validated questionnaire which measures the health status of patients with COPD, with a score ranging from 0 (no impairment) to 100 (worst possible health).
Mean change in HADS compared to MCID. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. MCID is the minimal clinically important difference for the validated tool. HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Mean change in modified BORG score compared to MCID. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. MCID is the minimal clinically important difference for the validated tool. The modified Borg scale is validated to assess breathlessness and is scored from 0 (not breathless) to 10 (maximal breathlessness).
Mean change in AKPS compared to MCID. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. MCID is the minimal clinically important difference for the validated tool. AKPS is a validated 10 point scale measuring performance status with 0 being normal health and 100 being dead.
Duration SGRQ score maintained above baseline. | 12 months
  To be measured in days. Within the whole longitudinal cohort and individual risk groups within the prognostic tools. SGRQ is a validated questionnaire which measures the health status of patients with COPD, with a score ranging from 0 (no impairment) to 100 (worst possible health).
Duration HADS score maintained above baseline. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. To be measured in days. HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Duration modified BORG score maintained above baseline. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. To be measured in days. The modified Borg scale is validated to assess breathlessness and is scored from 0 (not breathless) to 10 (maximal breathlessness).
Duration AKPS maintained above baseline. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools. To be measured in days. AKPS is a validated 10 point scale measuring performance status with 0 being normal health and 100 being dead.
Relation between clinically significant anxiety on discharge and survival. | 12 months
  As per the anxiety component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Relation between clinically significant depression on discharge and survival. | 12 months
  As per the depression component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Relation between clinically significant anxiety on discharge and quality of life. | 12 months
  As per the anxiety component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components. Quality of life as measured by the SGRQ, modified Borg and AKPS scores, with details of these scores described above.
Relation between clinically significant depression on discharge and quality of life. | 12 months
  As per the depression component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components. Quality of life as measured by the SGRQ, modified Borg and AKPS scores, with details of these scores described above.
Relation between clinically significant anxiety on discharge and functional status. | 12 months
  As per the anxiety component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components. Functional status as per the AKPS and SGRQ scores described above.
Relation between clinically significant depression on discharge and functional status. | 12 months
  As per the depression component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components. Functional status as per the AKPS and SGRQ scores described above.
Relation between clinically significant anxiety on discharge and readmissions. | 12 months
  As per the anxiety component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Relation between clinically significant depression on discharge and readmissions. | 12 months
  As per the depression component of the HADS tool - HADS is a validated questionnaire with a score range of 0 (healthy) to maximum 21 (abnormal) for both anxiety and depression components.
Best prognostic tool to predict poor QoL and/or death within one year, as per positive predictive value and sensitivity. | 12 months
  Within the whole longitudinal cohort and individual risk groups within the prognostic tools.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah M Gillespie, MBChB, Principal Investigator — Northumbria Healthcare NHS Foundation Trust
Locations (2):
- United Kingdom (2):
  - Newcastle Upon Tyne Hospitals NHS Foundation Trust, Newcastle upon Tyne, Tyne and Wear
  - Northumbria Healthcare NHS Foundation Trust, Cramlington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Echevarria C, Steer J, Heslop-Marshall K, Stenton SC, Hickey PM, Hughes R, Wijesinghe M, Harrison RN, Steen N, Simpson AJ, Gibson GJ, Bourke SC. The PEARL score predicts 90-day readmission or death after hospitalisation for acute exacerbation of COPD. Thorax. 2017 Aug;72(8):686-693. doi: 10.1136/thoraxjnl-2016-209298. Epub 2017 Feb 24. PMID 28235886
- [Background] Soler-Cataluna JJ, Martinez-Garcia MA, Sanchez LS, Tordera MP, Sanchez PR. Severe exacerbations and BODE index: two independent risk factors for death in male COPD patients. Respir Med. 2009 May;103(5):692-9. doi: 10.1016/j.rmed.2008.12.005. Epub 2009 Jan 7. PMID 19131231
- [Background] Thomas K et al. The GSF Prognostic Indicator Guidance. The Gold Standards Framework Centre in End of Life Care CIC; October 2011
- [Background] Almagro P, Soriano JB, Cabrera FJ, Boixeda R, Alonso-Ortiz MB, Barreiro B, Diez-Manglano J, Murio C, Heredia JL; Working Group on COPD, SpanishSociety of Internal Medicine*. Short- and medium-term prognosis in patients hospitalized for COPD exacerbation: the CODEX index. Chest. 2014 May;145(5):972-980. doi: 10.1378/chest.13-1328. PMID 24077342
- [Background] Puhan MA, Hansel NN, Sobradillo P, Enright P, Lange P, Hickson D, Menezes AM, ter Riet G, Held U, Domingo-Salvany A, Mosenifar Z, Anto JM, Moons KG, Kessels A, Garcia-Aymerich J; International COPD Cohorts Collaboration Working Group. Large-scale international validation of the ADO index in subjects with COPD: an individual subject data analysis of 10 cohorts. BMJ Open. 2012 Dec 12;2(6):e002152. doi: 10.1136/bmjopen-2012-002152. Print 2012. PMID 23242246
- [Background] Sundh J, Janson C, Lisspers K, Stallberg B, Montgomery S. The Dyspnoea, Obstruction, Smoking, Exacerbation (DOSE) index is predictive of mortality in COPD. Prim Care Respir J. 2012 Sep;21(3):295-301. doi: 10.4104/pcrj.2012.00054. PMID 22786813
- [Background] Highet G, Crawford D, Murray SA, Boyd K. Development and evaluation of the Supportive and Palliative Care Indicators Tool (SPICT): a mixed-methods study. BMJ Support Palliat Care. 2014 Sep;4(3):285-90. doi: 10.1136/bmjspcare-2013-000488. Epub 2013 Jul 25. PMID 24644193
- [Background] Steer J, Gibson J, Bourke SC. The DECAF Score: predicting hospital mortality in exacerbations of chronic obstructive pulmonary disease. Thorax. 2012 Nov;67(11):970-6. doi: 10.1136/thoraxjnl-2012-202103. Epub 2012 Aug 15. PMID 22895999
- [Background] Echevarria C, Steer J, Heslop-Marshall K, Stenton SC, Hickey PM, Hughes R, Wijesinghe M, Harrison RN, Steen N, Simpson AJ, Gibson GJ, Bourke SC. Validation of the DECAF score to predict hospital mortality in acute exacerbations of COPD. Thorax. 2016 Feb;71(2):133-40. doi: 10.1136/thoraxjnl-2015-207775. PMID 26769015
- [Background] Knaus WA, Wagner DP, Draper EA, Zimmerman JE, Bergner M, Bastos PG, Sirio CA, Murphy DJ, Lotring T, Damiano A, et al. The APACHE III prognostic system. Risk prediction of hospital mortality for critically ill hospitalized adults. Chest. 1991 Dec;100(6):1619-36. doi: 10.1378/chest.100.6.1619. PMID 1959406
- [Background] Meguro M, Barley EA, Spencer S, Jones PW. Development and Validation of an Improved, COPD-Specific Version of the St. George Respiratory Questionnaire. Chest. 2007 Aug;132(2):456-63. doi: 10.1378/chest.06-0702. Epub 2007 Jul 23. PMID 17646240
- [Background] Zigmond AS, Snaith RP. The hospital anxiety and depression scale. Acta Psychiatr Scand. 1983 Jun;67(6):361-70. doi: 10.1111/j.1600-0447.1983.tb09716.x. PMID 6880820
- [Background] Abernethy AP, Shelby-James T, Fazekas BS, Woods D, Currow DC. The Australia-modified Karnofsky Performance Status (AKPS) scale: a revised scale for contemporary palliative care clinical practice [ISRCTN81117481]. BMC Palliat Care. 2005 Nov 12;4:7. doi: 10.1186/1472-684X-4-7. PMID 16283937
- [Background] Steer J, Norman EM, Afolabi OA, Gibson GJ, Bourke SC. Dyspnoea severity and pneumonia as predictors of in-hospital mortality and early readmission in acute exacerbations of COPD. Thorax. 2012 Feb;67(2):117-21. doi: 10.1136/thoraxjnl-2011-200332. Epub 2011 Sep 6. PMID 21896712
- [Background] Kendrick KR, Baxi SC, Smith RM. Usefulness of the modified 0-10 Borg scale in assessing the degree of dyspnea in patients with COPD and asthma. J Emerg Nurs. 2000 Jun;26(3):216-22. doi: 10.1016/s0099-1767(00)90093-x. PMID 10839848

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/21/NCT03657121/Prot_SAP_001.pdf